CLINICAL TRIAL: NCT06606366
Title: Study on the Contribution of the Genetic Tumor Profile Obtained by Circulating Tumor DNA Analysis in the Multidisciplinary Molecular Biology Meeting of Eastern PACA
Acronym: TARGET
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Antoine Lacassagne (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2020/58; 2024-A01332-45 (Other: ANSM)
Record Dates: First submitted 2024-09-18; First posted 2024-09-23 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Neoplasm Malignant
Keywords: Liquid biopsy
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Experimental (Experimental): For this study, the included patients will have a blood sample (36 mL) taken. Molecular analyses will be performed on this blood sample (liquid biopsy) in addition to the molecular analyses routinely conducted on the tumor sample (solid biopsy).
  Interventions: Procedure: Blood sample taken for the liquid biopsy

INTERVENTIONS:
Procedure: Blood sample taken for the liquid biopsy — 36 mL will be taken for the study.

SUMMARY:
This study will evaluate the diagnostic performance of liquid biopsy for identifying molecular abnormalities among patients managed by the Multidisciplinary Molecular Biology Meeting. The gold standard considered in this study is the solid biopsy.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old.
* Advanced-stage malignant solid tumor managed in a non-curative context.
* Patient eligible for Multidisciplinary molecular biology meeting with available archived tumor material (frozen or FFPE block, less than 5 years old) or a biopsiable tumor lesion.
* Performance status of 0 or 1.
* Patient able to read, write, and understand the French language.
* Patient has read the information sheet and signed the informed consent.
* Patient has social security coverage.

Exclusion Criteria:

* Previous or concurrent cancer diagnosed or treated within the last 5 years, except for in situ carcinoma of the cervix, basal cell or squamous cell carcinoma of the skin, and adequately treated in situ carcinoma of the bladder.
* Severe or uncontrolled systemic disease.
* Any condition which, in the investigator's judgment (geographical, social, or psychological factors, etc.), makes the patient unable to comply with study follow-up and procedures.
* Patient considered a vulnerable person; vulnerable persons are defined in Articles L1121-5 to L1121-8:

  * Pregnant women, women in labor, and breastfeeding mothers,
  * Persons deprived of liberty by judicial or administrative decision, individuals hospitalized without consent under Articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of Article L. 1121-8,
  * Persons admitted to a healthcare or social institution for reasons other than research,
  * Adults unable to give their consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Estimated)
Dates: Start 2025-03-03 (Actual); Primary Completion 2027-06-03 (Estimated); Study Completion 2027-06-03 (Estimated)

PRIMARY OUTCOMES:
Sensitivity of liquid biopsy versus solid biopsy (gold standard) | 1 month
  The primary endpoind is the sensitivity of liquid biopsy versus solid biopsy as the gold standard for detecting genomic alterations evaluated in the studied gene panel.
  The panel will consist of 70 genes common to the PanoraMix panels (125 genes, FFPE) and Avida (104 genes, cpDNA).

SECONDARY OUTCOMES:
Specificity of liquid biopsy versus solid biopsy (gold standard) | 1 month
  The specificity of liquid biopsy versus solid biopsy as the gold standard in the detection of genomic alterations evaluated in the studied gene panel.
Failure rate of molecular screening | 1 month
  The failure rate of molecular screening (defined as the inability to provide the genetic profile from the liquid biopsy due to technical failure).
Clinical factors predictive of the sensitivity of liquid biopsy. | 1 month
  Clinical factors predictive of the sensitivity of liquid biopsy.
Rate of unexploitable results | 1 month
  The rate of unexploitable results, defined as the rate of results that do not allow for classification for each technique of the results as True Positive, False Positive, False Negative, or True Negative.
Time required to obtain each analysis | 1 month
  The time required to obtain each analysis, defined as the time between the prescription of the test and the delivery of the result.

CONTACTS AND LOCATIONS:
Locations (1):
- Centre Antoine Lacassagne, Nice, France

IPD SHARING:
Plan to Share IPD: Undecided